CLINICAL TRIAL: NCT05259397
Title: A PHASE 1, OPEN-LABEL, DOSE ESCALATION AND EXPANSION STUDY OF PF-07225570 EITHER ALONE OR IN COMBINATION WITH AN ANTI-PD-1 ANTIBODY, IN PARTICIPANTS WITH RECURRENT NON-MUSCLE INVASIVE BLADDER CANCER
Brief Title: PF-07225570 Alone or in Combination With an Anti-PD-1 Antibody in Recurrent Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pfizer has decided to terminate Study C4661001 due to strategic considerations. This decision is not due to any specific safety reasons or requests from any regulatory authorities. No participants have been enrolled in this study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4661001; 2021-005858-28 (EudraCT Number)
Record Dates: First submitted 2022-02-15; First posted 2022-02-28 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Bladder Cancer
Keywords: Recurrent Non-Muscle Invasive Bladder Cancer (NMIBC); Urothelial cancer; Toll-like receptor 7 (TLR7); Toll-like receptor 8 (TLR8)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Antibodies

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1A PF-07225570 monotherapy (Experimental): Intravesical (IVe) Single Agent Dose Escalation
  Interventions: Drug: PF-07225570
- Part 1B PF-07225570 and sasanlimab (Experimental): PF-07225570 IVe and sasanlimab Subcutaneous (SQ) Combination Dose Escalation
  Interventions: Drug: PF-07225570; Drug: sasanlimab
- Part 2A PF-07225570 monotherapy (Experimental): IVe Single Agent Dose Expansion
  Interventions: Drug: PF-07225570
- Part 2B PF-07225570 and sasanlimab (Experimental): PF-07225570 IVe and sasanlimab SQ Combination Dose Expansion
  Interventions: Drug: PF-07225570; Drug: sasanlimab

INTERVENTIONS:
Drug: PF-07225570 — PF-07225570 given IVe in a 28-day cycle (as induction and maintenance regimen). Multiple dose levels will be evaluated.
Drug: sasanlimab — Sasanlimab will be administered SQ on day 1 of each 28 day cycle.
  Other Names: anti-PD-1 (programmed cell death protein-1) antibody
  Arms: Part 1B PF-07225570 and sasanlimab; Part 2B PF-07225570 and sasanlimab

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of PF-07225570 alone or in combination with an anti-PD-1 antibody in participants with recurrent non-muscle invasive bladder cancer. This study consists of 2 parts, single agent dose escalation (Part 1A), dose finding of PF-07225570 in combination with anti-PD-1 antibody (Part 1B) and dose expansion (Part 2).

ELIGIBILITY:
Inclusion Criteria:

Histological confirmed and documented diagnosis of non-muscle invasive urothelial carcinoma

Participants with recurrent non-muscle invasive bladder cancer (intermediate risk or high risk)

Ineligible for or elected not to undergo radical cystectomy

No evidence of upper tract urothelial cancer or cancer within the prostatic urethra as documented by imaging studies performed within 6 months of enrollment

Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1

Adequate bone marrow, renal and liver function

Exclusion Criteria:

Evidence of muscle-invasive, locally advanced or metastatic urothelial carcinoma or concurrent extravesical, non-muscle invasive urothelial carcinoma

Macroscopic hematuria, traumatic catheterization or active urinary tract infection

Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent

Active, uncontrolled bacterial, fungal, or viral infection, including (but not limited to) Hepatitis B, Hepatitis C, and known Human Immunodeficiency Virus infection or Acquired Immunodeficiency Syndrome-related illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose limiting toxicities | Baseline up to 28 days
Number of Participants with Adverse Events (AEs) according to Severity | Baseline up to approximately 24 months
Number of Participants with AEs according to Seriousness | Baseline up to approximately 24 months
Number of Participants with AEs according to Relationship | Baseline up to approximately 24 months

SECONDARY OUTCOMES:
Proportion of participants with carcinoma in situ (CIS) achieving complete response at any time after first dose of PF 07225570 | Baseline up to 24 months
Durability of complete responses (CRs) as measured from time of documented CR to time of high-grade tumor recurrence, disease progression, or death (whichever occurs first) in participants who achieved a CR | Baseline up to 24 months
For participants with high-grade Ta/ T1 disease only, Proportion of participants without high-grade-recurrence at each assessment visit. | Baseline up to 24 months
  Ta is defined as the stage of bladder cancer as a non-invasive papillary carcinoma. T1 is defined as the stage of cancer in which the cancer cells are only growing in the most superficial layer of tissues and have not grown into deeper tissues; in bladder cancer, T1 is defined as an invasion into the lamina propria without invasion into the muscularis propria
Maximum Observed Plasma Concentration (Cmax) of PF-7225570 after a single dose | Pre-dose on Cycle 1 (each cycle is 28 days) Day 1 and at 0.5, 1, 2, 3, 4, 6 and 24 hours after instillation
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07225570 after a single dose | Pre-dose on Cycle 1 (each cycle is 28 days) Day 1 and at 0.5, 1, 2, 3, 4, 6 and 24 hours after instillation
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-07225570 after a single dose | Pre-dose on Cycle 1 (each cycle is 28 days) Day 1 and at 0.5, 1, 2, 3, 4, 6 and 24 hours after instillation
Concentration from maximum to steady state (Cmax,ss) of PF-07225570 after multiple doses | Pre-dose on Cycle 1 (each cycle is 28 days) Day 1 and at 2 hours after instillation
Time from maximum concentration to steady state (Tmax,ss) of PF-07225570 after multiple doses | Pre-dose on Cycle 1 (each cycle is 28 days) Day 1 and at 2 hours after instillation
Area under the curve from specified time to steady state (AUCτ,ss) of PF-07225570 after multiple doses | Pre-dose on Cycle 1 (each cycle is 28 days) Day 1 and at 2 hours after instillation
Urine PF-07225570 concentration after a single dose | Pre-dose on Cycle 1 (each cycle is 28 days) Day 1 and at 0-2 hours, and 4 - 6 hours post-instillation on Cycle 1 Day 1
Urine PF-07225570 concentration after multiple doses | Pre-dose on Cycle 1 (each cycle is 28 days) Day 1 and at 0-2 hours and 2 - 4 hours post-instillation.
Progression-Free Survival | Baseline up to 24 months
Incidence of Radical Cystectomy | Baseline up to 24 months
Overall survival | Baseline up to 3 years
Serum sasanlimab concentrations | Pre-dose (within 6 hours) before each administration
Incidence and titers of neutralizing antibodies (NAb) against sasanlimab | Pre-dose (within 6 hours) before each administration
Incidence and titers of anti-drug antibodies (ADA) against sasanlimab | Pre-dose (within 6 hours) before each administration

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (2):
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - CUMC Research Pharmacy, New York, New York
- Poland (2):
  - Szpital Specjalistyczny im. Sw. Rodziny SPZOZ, Warsaw
  - Medical Concierge Centrum Medyczne, Warsaw

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4661001